CLINICAL TRIAL: NCT03118232
Title: Project PROTECT: Protecting Nursing Homes From Infections and Hospitalization
Acronym: PROTECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); University of Massachusetts, Amherst (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Huang, Professor and Medical Director of Epidemiology and Infection Prevention, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20151805
Record Dates: First submitted 2017-02-21; First posted 2017-04-18 (Actual); Results first posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Hospitalization; Infection
Keywords: Nursing Homes; Health Facilities; Infections; Readmissions; Multi-Drug resistance; Antibiotic Use
MeSH Terms: conditions — Infections | interventions — chlorhexidine gluconate; Iodophors; Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Decolonization (Active Comparator): Nursing homes assigned to this arm will perform decolonization using topical antiseptic products.
  Interventions: Drug: Chlorhexidine gluconate (CHG); Drug: Iodophor (10% povidone-iodine)
- Routine Bathing (No Intervention): Routine bathing per facility protocol.

INTERVENTIONS:
Drug: Chlorhexidine gluconate (CHG) — 2% no-rinse chlorhexidine gluconate (CHG) for bed bathing and 4% rinse-off CHG showering. Bathing frequency will be per routine plus admission bathing.
  Arms: Decolonization
Drug: Iodophor (10% povidone-iodine) — Nasal decolonization using topical 10% povidone-iodine nasal swabs will be applied to all residents on admission for 5 days twice daily plus every other week Monday-Friday using a twice daily regimen.
  Arms: Decolonization

SUMMARY:
This is a cluster-randomized trial of nursing homes to assess whether decolonization with routine chlorhexidine bathing and periodic use of nasal antiseptics can reduce hospitalizations associated with infections, antibiotic utilization, and multi-drug resistant organism (MDRO) prevalence. The comparator arm will be routine bathing care.

ELIGIBILITY:
Inclusion Criteria

Nursing homes will be eligible to participate if they meet the following criteria:

* Licensed nursing home in Orange County or Southern Los Angeles County serving adults
* Minimal use of chlorhexidine bathing*
* Minimal use of nasal decolonization* *Minimal use defined as <15% of residents receiving at least one chlorhexidine bath or nasal decolonization treatment during their nursing home stay.

Exclusion Criteria

Nursing homes will not be eligible to participate if they meet the following criteria:

* Facilities routinely using decolonization
* Dedicated psychiatric nursing homes
* Facilities with a resident population with >=20% combative patients
* Pediatric facilities

Note: in any participating nursing home, residents with active end-of-life comfort care only measures are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13952 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Huang, MD MPH, Principal Investigator — University of California, Irvine; Loren Miller, MD MPH, Study Director — Harbor UCLA; James McKinnell, MD, Study Director — Harbor UCLA
Locations (28):
- United States (28):
  - Buena Vista Care Center, Anaheim, California
  - Walnut Village Rehabilitation and Care Center, Anaheim, California
  - Anaheim Crest Nursing Center, Anaheim, California
  - Sun Mar Nursing Center, Anaheim, California
  - West Anaheim Extended Care, Anaheim, California
  - Bel Tooren Villa Convalescent Hospital, Bellflower, California
  - Capistrano Beach Care Center, Capistrano Beach, California
  - Downey Care Center, Downey, California
  - Gordon Lane Care Center, Fullerton, California
  - Windsor Gardens Care Center of Fullerton, Fullerton, California
  - Terrace View Care Center, Fullerton, California
  - Pacific Haven Subacute Healthcare Center, Garden Grove, California
  - Las Flores Convalescent Hospital, Gardena, California
  - Park Regency Care Center, La Habra, California
  - Regency Oaks Post Acute Care Center, Long Beach, California
  - Windsor Convalescent of North Long Beach, Long Beach, California
  - Bixby Knolls Healthcare Center, Long Beach, California
  - Pacific Villa Inc., Long Beach, California
  - Vista Cove Care Center at Long Beach, Long Beach, California
  - Intercommunity Care Center, Long Beach, California
  - Royal Oaks Care Center, Lynwood, California
  - Norwalk Skilled Nursing and Wellness Center, Norwalk, California
  - Villa Elena Care Center, Norwalk, California
  - Harbor Post-Acute Care Center, Torrance, California
  - Heritage Rehabilitation Center, Torrance, California
  - Sunnyside Nursing Center, Torrance, California
  - Torrance Care Center West, Torrance, California
  - Del Amo Gardens Care Center, Torrance, California

IPD SHARING:
Plan to Share IPD: No
The resource sharing plan involves sharing 1) sharing of trial materials and tools, and 2) making bacterial isolates available.

REFERENCES:
- [Derived] Miller LG, McKinnell JA, Singh RD, Gussin GM, Kleinman K, Saavedra R, Mendez J, Catuna TD, Felix J, Chang J, Heim L, Franco R, Tjoa T, Stone ND, Steinberg K, Beecham N, Montgomery J, Walters D, Park S, Tam S, Gohil SK, Robinson PA, Estevez M, Lewis B, Shimabukuro JA, Tchakalian G, Miner A, Torres C, Evans KD, Bittencourt CE, He J, Lee E, Nedelcu C, Lu J, Agrawal S, Sturdevant SG, Peterson E, Huang SS. Decolonization in Nursing Homes to Prevent Infection and Hospitalization. N Engl J Med. 2023 Nov 9;389(19):1766-1777. doi: 10.1056/NEJMoa2215254. Epub 2023 Oct 10. PMID 37815935

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Nursing Homes
Period: Overall Study
Arm/Group | Decolonization | Routine Bathing
Started | 7388; 14 Nursing Homes | 6564; 14 Nursing Homes
Completed | 7388; 14 Nursing Homes | 6564; 14 Nursing Homes
Not Completed | 0; 0 Nursing Homes | 0; 0 Nursing Homes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decolonization | Routine Bathing | Total
Number analyzed (Participants) | 7388 | 6564 | 13952
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.7 (4.2) | 76.6 (5.8) | 76.2 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4180 | 3602 | 7782
  Male | 3208 | 2962 | 6170
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1042 | 1312 | 2354
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 841 | 1042 | 1883
  White | 3749 | 2666 | 6415
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1756 | 1544 | 3300
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7388 | 6564 | 13952

OUTCOME MEASURES:

1. Primary Outcome: Hospital Transfers Due to Infection
Description: Probability that a transfer to a hospital is due to an infection
Time Frame: 18 months
Population: Analysis is of residents accounting for clustering in 28 nursing homes
Measure: Number; unit: Transfers
Arm/Group | Decolonization | Routine Bathing
Number analyzed (Participants) | 7388 | 6564
Transfers | 1243 | 1780
Statistical Analysis 1: Comparison: Decolonization vs Routine Bathing; Test type: Other — The risk ratios reflect the risk of transfer to a hospital during the intervention period relative to the baseline period in each trial group; p < 0.001, Mixed Models Analysis; Difference in Risk Ratio = 16.6, 95% CI 2-sided [11.0 to 21.8]

2. Secondary Outcome: All Hospital Transfers
Description: Probability that a discharge is to a hospital
Time Frame: 18 months
Population: Analysis is of residents accounting for clustering in 28 nursing homes
Measure: Number; unit: Transfers
Arm/Group | Decolonization | Routine Bathing
Number analyzed (Participants) | 7388 | 6564
Transfers | 2388 | 2857
Statistical Analysis 1: Comparison: Decolonization vs Routine Bathing; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Difference in Risk Ratio = 14.6, 95% CI 2-sided [9.7 to 19.2]

3. Other Pre Specified Outcome: Multidrug-resistant Organism (MDRO) Colonization (Secondary Manuscript)
Description: Probability of colonization with any multidrug-resistant organism (MDRO): (MRSA, VRE, ESBL, CRE)
Time Frame: Once in baseline and once at end-intervention (month 15-18 of intervention period)
Measure: Count of Participants; unit: Participants
Arm/Group | Decolonization | Routine Bathing
Number analyzed (Participants) | 550 | 650
Participants | 176 | 307

4. Other Pre Specified Outcome: Hospital Transfers Due to Infection in Long Stay and Short Stay Subsets (Secondary Manuscript, Added by Steering Committee Decision on 3/22/2017)
Description: Probability that a transfer to a hospital is due to an infection for long stay and short stay resident subsets
Time Frame: 18 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: All Hospital Transfers in Long Stay and Short Stay Subsets (Secondary Manuscript, Added by Steering Committee Decision on 3/22/2017)
Description: Probability that a discharge is to a hospital for long stay and short stay resident subsets
Time Frame: 18 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Emergency Department Transfers Due to Infection (Secondary Manuscript, Added by Steering Committee Decision on 3/22/2017)
Description: Probability that a resident is sent to the emergency department for an infection, overall for long stay and short stay resident subsets
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Decolonization | Routine Bathing
All-Cause Mortality (participants affected / at risk) | 0/7388 | 0/6564
Serious Adverse Events (participants affected / at risk) | 0/7388 | 0/6564
Other Adverse Events (participants affected / at risk) | 35/7388 | 0/6564
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decolonization (N=7388) | Routine Bathing (N=6564)
Rashes (Product Issues) | 34 (34) | 0 (0)
Sore throat (Product Issues) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT03118232/Prot_SAP_000.pdf